CLINICAL TRIAL: NCT02781870
Title: Randomized Single-center Study on Laparoscopic Groin Hernia Repair by a 3D ENDOLAP Visible With and Without LiquiBand Fix 8 Mesh Fixation
Brief Title: Laparoscopic Groin Hernia Repair by a 3D ENDOLAP Visible Mesh With or Without LiquiBand Fix 8 Mesh Fixation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Collaborators: Duomed (Industry)
Responsible Party: Principal Investigator, Filip Muysoms, abdominal wall surgeon, Algemeen Ziekenhuis Maria Middelares
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: EUGENE STUDY
Record Dates: First submitted 2016-05-10; First posted 2016-05-25 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Hernia; Recurrence
MeSH Terms: conditions — Hernia; Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No-fixation (Other): These patients will be randomized during the operation, at the time of mesh placement to receive the 3D ENDOLAP visible without fixation.
  Interventions: Procedure: No-fixation
- LiquiBand Fix glue fixation (Experimental): These patients will be randomized during the operation, at the time of mesh placement to receive the 3D ENDOLAP visible with LiquiBand® Fix 8™ glue fixation.
  Patients will be operated in a standard procedure to receive the 3D ENDOLAP visible with LiquiBand® Fix 8™ glue fixation.
  Interventions: Procedure: LiquiBand Fix8 glue fixation

INTERVENTIONS:
Procedure: LiquiBand Fix8 glue fixation — Patients will be operated in a standard procedure to receive the 3D ENDOLAP visible with LiquiBand® Fix 8™ glue fixation.
  Other Names: LiquiBand Fix8 glue
  Arms: LiquiBand Fix glue fixation
Procedure: No-fixation — Patients will be operated in a standard procedure to receive the 3D ENDOLAP visible without glue fixation.
  Arms: No-fixation

SUMMARY:
This study aims to visualize the implanted mesh in vivo by MRI in 20 patients at 1 month and 12 months post-operatively. Moreover, we want to evaluate the safety and efficiency of non-penetration mesh fixation techniques using pre-designed ENDOLAP 3D visible mesh placement versus mesh fixation using a synthetic LiquiBand Fix 8 glue for laparoscopic treatment of groin hernias.

A total of 100 male and female patients will be entered in the trial in Maria Middelares Ghent, for which an inclusion period of 24 months is anticipated. Four surgeons of the department of surgery will screen all eligible consecutive patients for inclusion in the study. They will inform all patients about the surgery and the follow-up with MRI scan thereafter.

DETAILED DESCRIPTION:
Inguinal hernia is a common disease with a high lifetime risk; 27 % for men and 3% for women. These hernias can be categorized as lateral, medial or femoral according to the classification of the European Hernia Society. The manifestations may vary from an asymptomatic swelling till an incarcerated or strangulated hernia requiring an urgent operation.

The introduction of mesh reinforcement for groin hernia repair has resulted in reducing the rate of recurrences and chronic pain. Moreover, laparoscopic repair techniques made it possible to place the mesh in de pre-peritoneal space by a transperitoneal (TAPP) or pre-peritoneal (TEP) approach. These minimally invasive techniques are not only associated with less chronic pain of numbness, but also with an earlier return to normal activities or work. A favor for one of the two techniques has not yet been proven.

Also, the repair of groin hernias always goes along with a discussion about placing the optimal mesh, the optimum mesh size and the optimal fixation method of the mesh. There are a lot of meshes available of different materials, in different sizes and with different properties.

The majority of all meshed need to be fixed to the abdominal wall. Meshes as the anatomic ProGrip Laparoscopic self-fixating mesh (Covidien) has been developed with self-fixating properties due to the polylactic acid micro-grips on one side of the mesh which secures the mesh without requiring any other form of fixation. While the ENDOLAP 3D visible mesh (Dynamesh) has been developed with a pre-shaped form that fits the defect naturally and therefore makes a fixation redundant.

However, no consensus on the best method of mesh fixation or even non-fixation can be found in the common literature. Penetrating fixation methods of the mesh have a strong positioning as result, but for inguinal hernia, mesh fixation using titanium tacks with or without sutures clearly indicated more development of postoperative pain and discomfort for the patient. Current recommendations are to avoid penetrating fixation and replace this by either no fixation or fixation with glue. This will decrease pain but should not risk a less stable mesh fixation ongoing with recurrence due to mesh shifting of mesh shrinkage. It is known that the majority of implanted meshes shrink to an extent, which might be of disadvantage for the patient. This has already been demonstrated in several animal studies, but clinical information on the mesh shrinkage is rare and mostly a result from revisional surgery.

LiquiBand Fix 8 glue is a new, innovative hernia mesh fixation device providing strong and secure mesh fixation without causing any tissue damage or mechanical trauma. LiquiBand Fix 8 received CE mark approval in May 2014.

All ordinary meshes for groin hernia repair, based on polymeric textile, are invisible to conventional imaging techniques, inclusive "magnetic resonance imaging" (MRI). The ENDOLAP 3D mesh visible (Dynamesh), developed by a unique method, contains an amount of iron particles, woven in the ordinary structure of the mesh, which allows an imaging in the MRI.

ELIGIBILITY:
Inclusion Criteria:

* adult patients presenting with primary unilateral inguinal hernia
* patients planed for a laparoscopic repair

Exclusion Criteria:

* Age below 18 years
* recurrent or incarcerated hernias
* open hernia repair and bilateral hernias
* concomitant repair of another kind of abdominal hernia
* combined surgical procedures
* no informed consent
* pregnant women
* ASA score 4 or more
* contra-indications for MRI scans.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
visualization of mesh surface | 12 months
  Visualization of the mesh surface at 12 months postoperative observed with MRI scan rate after laparoscopic repair of unilateral inguinal hernias using the 3D-Endolap visible mesh with or without LiquiBand® Fix 8™ glue fixation.

SECONDARY OUTCOMES:
visualization of mesh surface | 1 month
  Visualization of the mesh surface at 1 month postoperative observed with MRI scan
recurrence of inguinal hernia | 1 month, 12 months, 36 months and 60 months
  Recurrence rate of inguinal hernia measured at 1 month, 12, 36 and 60 months clinically of by ultrasound as indicated.

OTHER OUTCOMES:
Quality of Life assessment | 1 month, 12 months, 36 months and 60 months
  Quality of Life assessment with the EuraHS QoL

CONTACTS AND LOCATIONS:
Overall Officials: Filip Muysoms, MD, PhD, Principal Investigator — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ Maria Middelares, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mayer F, Niebuhr H, Lechner M, Dinnewitzer A, Kohler G, Hukauf M, Fortelny RH, Bittner R, Kockerling F. When is mesh fixation in TAPP-repair of primary inguinal hernia repair necessary? The register-based analysis of 11,230 cases. Surg Endosc. 2016 Oct;30(10):4363-71. doi: 10.1007/s00464-016-4754-8. Epub 2016 Feb 17. PMID 26886454
- [Background] Klobusicky P, Feyerherd P. Innovation in Laparoscopic Inguinal Hernia Reparation - Initial Experiences with the Parietex Progrip Laparoscopic() - Mesh. Front Surg. 2015 Jun 25;2:28. doi: 10.3389/fsurg.2015.00028. eCollection 2015. PMID 26161386